CLINICAL TRIAL: NCT04387825
Title: Lipograft Safety Enriched With Vascular Stromal Fraction Derived From Adipose Tissue, to Treatment of Digital Joint Fibrosis and Refractory Ischemic Digital Ulcers Caused by Systemic Sclerosis
Brief Title: Safety Of Fat Micrografts With Adipose-Derived Stromal Vascular Fraction In Hands Of Patients With Systemic Sclerosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Collaborators: National Council of Science and Technology, Mexico (Other)
Responsible Party: Principal Investigator, Martín Iglesias, Plastic Surgeon, Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCI-1505-15/15-1; 290250 (Other Grant/Funding Number: CONACYT)
Record Dates: First submitted 2020-05-10; First posted 2020-05-14 (Actual); Last update posted 2020-05-15 (Actual); Status verified 2020-05

CONDITIONS: Systemic Sclerosis
Keywords: Hand deformities in Systemic sclerosis
MeSH Terms: conditions — Scleroderma, Systemic

STUDY DESIGN:
Intervention Model Description: Adipose Derived Stromal Vascular Fraction (ADSVF) was obtained in a laboratory by enzymatic digestion of fat graft harvested by liposuction. This ADSVF and micro fat grafts were applied into the hands with fibrosis and digital ulcers caused by Systemic Sclerosis in the experimental group. The control group was treated with medical treatment only
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group (Experimental): 40 ml of fat was mixed with 2 ml of ADSVF and placed in 1-ml and 3-ml syringes. Using a 19-gauge blunt cannula (0.8 mm), 0.5 ml was applied to the radial and ulnar edge of each metacarpal phalangeal (MP) and interphalangeal (IP) joint in contact with each neurovascular digital pedicle and 3 ml was applied to each side of the metacarpal trapezius joint, together with 10 ml distributed subcutaneously throughout the palm of the hand and 10 ml evenly distributed on the back of the hand
  Interventions: Drug: ADSVF application in the right hand
- Control (No Intervention): Evolution and medical therapy effects were observed in the control group.

INTERVENTIONS:
Drug: ADSVF application in the right hand — 40 ml of fat was mixed with 2 ml of ADSVF and placed in 1-ml and 3-ml syringes. Using a 19-gauge blunt cannula (0.8 mm), 0.5 ml was applied to the radial and ulnar edge of each metacarpal phalangeal (MP) and interphalangeal (IP) joint in contact with each neurovascular digital pedicle and 3 ml was applied to each side of the metacarpal trapezius joint, together with 10 ml distributed subcutaneously throughout the palm of the hand and 10 ml evenly distributed on the back of the hand
  Other Names: Medical treatment
  Arms: Experimental group

SUMMARY:
Systemic sclerosis (SS) causes microvascular alteration in the hand and subsequently pain, skin fibrosis, and osteoarticular deformities. These injuries initiate functional decline of the hand and decrease patient quality of life.

Local application of adipose-derived stromal vascular fraction (ADSVF) has been proposed as an emerging treatment. There are reports about the good results obtained after ADSVF treatment in this kind of patients. For these reasons , we aimed to evaluate the safety and clinical effect of application of fat micrografts enriched with ADSVF to the hands of patients with SS.

DETAILED DESCRIPTION:
The regenerative properties of adipose stem cells (ASCs) existing in the mixed cell fraction obtained by enzymatic digestion of adipose tissue, termed adipose-derived stromal vascular fraction (ADSVF), were initially described in 2002. These cells have the characteristics of being multipotent and exerting local angiogenic, anti-inflammatory, antifibrotic, immunomodulatory, and regenerative effects after application. ASCs express their angiogenic properties most effectively in a hypoxic environment.

For the above reasons, and because of its abundance in fat, easy acquisition, and almost immediate availability for use, ADSVF has positioned itself as an alternative for repair and regeneration of ischemic tissue.

Application of decanted fat, centrifuged fat, and ADSVF, has consistently and significantly improved pain, Raynaund Phenomen, and healing of digital ulcers in the hands of patients with SS, and thus improved their quality of life. Other inconsistent benefits have also been reported, such as decreased digital circumference, improvement in digital mobility and strength, improvement in formation of new subungual capillaries, and improvement in function through evaluation of the Cochin scale.

Based on the above findings, and because changes in the hands of patients with SS may arise through loss of adipocytes and defective stem cell function, we designed the present study with the aim of evaluating the safety, reproducibility, and clinical effects of application of fat micrografts enriched with ADSVF to the hands of patients affected with SS in a controlled clinical trial.

The experimental and control groups each contained 10 patients diagnosed with SS according to the criteria of the American College of Rheumatology and the LeRoy-Medsger criteria.

It was decided to carry out the treatment on the most affected hand of the patients, which was the right hand in the entire experimental group. ADSVF-enriched fat micrografts were applied to the experimental group. Evolution and medical therapy effects were observed in the control group.

The fat was obtained by liposucction and the ADSVF was processed in laboratory.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with SS, according to the criteria of the American College of Rheumatology and those of LeRoy-Medsger.
* Over 18 years old,
* BMI> 18 kg / m2.
* Patients received stable vasoactive and immunosuppressive therapies, for at least 1 month before being enrolled in the study, and this was continued unchanged throughout the study.

Exclusion Criteria:

* infected digital ulcers
* comorbidities that could affect hand function
* alcoholism
* drug abuse
* history of family cancer
* Patients with hyperbaric therapy one month before
* Botulinum toxin one month before
* surgical sympathectomy one month before

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-08-13 (Actual); Primary Completion 2019-05 (Actual); Study Completion 2020-05 (Actual)

PRIMARY OUTCOMES:
Pain before the treatment and every day during one week after the treatment, and each 28 days after de first week until the 168 day | 168 days
  Evaluation with Numerical Pain Rating Scale(NPRS) before, and after the intervention. The minimum value is 0 and maximum is 10. High value is worst
Frequency of Raynaud Phenomenon | 168 days
  Frequency, number of events per day/week;
Duration of Raynaud Phenomenon | 168 days
  Duration of minutes in every event.

SECONDARY OUTCOMES:
Digital Total active Motion | 168 days
  Goniometry, kapandjy Test
Digital oximetry | 168 days
  Transcutaneous Oximetry
Digital Ulcers | 168 days
  Number of ulcers
Health status and disability index | 168 days
  Evaluated by Sclerosis Health assessment Questionnarie (SHAQ) scale, before and at the end of the study. The value are from 0 to 3. A result >1.25 is worst
Hand Function | 168 days
  Cochin Scale, the values are from 0 to 90, higher values means poor function
Health-related quality of life, before de treatment and at the end of the study | 168 days
  Short Form 36 (SF-36) scale. High values is poor patient health
Vascularity of the nail bed | 168 days
  Videocapillaroscopy by field
Skin affection of the hand | 168 days
  Modified Rodnan scale, the values are from 0 to 51. High values higher skin fibrosis

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Hinojosa, MD, Study Chair — Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Locations (1):
- Instituto Nacional de Ciencias Medicas y Nutricion salvador Zubiran, México, Mexico

IPD SHARING:
Plan to Share IPD: No